CLINICAL TRIAL: NCT05151614
Title: Adjuvant Use Of Colchicine With The Standard Therapy In Moderate And Severe Corona Virus Disease-19 Infection: Randomized Controlled Clinical Trial
Brief Title: Adjuvant Use Of Colchicine With The Standard Therapy In Moderate And Severe Corona Virus Disease-19 Infection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Faiq Gorial, Professor, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRO21230003
Record Dates: First submitted 2021-11-27; First posted 2021-12-09 (Actual); Last update posted 2021-12-09 (Actual); Status verified 2021-11

CONDITIONS: COVID-19 Pandemic
MeSH Terms: conditions — COVID-19 | interventions — Colchicine

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Colchicine group (Experimental): Colchicine 0.5 mg tab 1x2 for 1 week then o.5mg tab. 1x1 for another week + the standard therapy
  Interventions: Drug: Colchicine 0.5 MG
- Control group (No Intervention): The patients in this group will receive only standard care which will include all or some of the following, according to the clinical condition of each patient:
  * Acetaminophen 500mg on need
  * Vitamin C 1000mg twice/ day
  * Zinc 75-125 mg/day
  * Vitamin D3 5000IU/day
  * Azithromycin 250mg/day for 5 days
  * Oxygen therapy/ C-Pap if needed
  * Dexamethasone 6 mg/day or methylprednisolone 40mg twice per day, if needed
  * Mechanical ventilation, if needed

INTERVENTIONS:
Drug: Colchicine 0.5 MG — Colchicine 0.5 mg tab 1x2 for 1 week then o.5mg tab. 1x1 for another week + the standard therapy ( total duration of colchicine 14 days).
  Other Names: Colchicine
  Arms: Colchicine group

SUMMARY:
The study included 2 arms Colchicine group: Colchicine + standard therapy of COVID-19 Control group: Standard therapy of COVID-19

DETAILED DESCRIPTION:
This study will be a randomized controlled trial with 2 arms study trial 1:1 allocation. The sample size was calculated and we need a total of 160 patients (80 Colchicine add on group and 80 controls)

ELIGIBILITY:
Inclusion Criteria:

* 1. Patients with age above 18 years and of any gender 2. Definite diagnosis of COVID-19 according to the WHO classification criteria 3. Patients symptomatic for no more than three days for mild-moderate cases, no more than two days after being severe cases 4. Understands and agrees to comply with planned study procedures.

Exclusion Criteria:

1. Patients refuse to enrol in the study
2. Patients with hypersensitivity to colchicine
3. Patients with chronic diseases: Renal failure with eGFR<30 ml/min; chronic liver disease with hepatic failure (AST/ALT > 3x normal).; decompensated heart failure, long QT syndrome (QTc >450 msec.), and uncontrolled arrhythmia; inflammatory bowel disease, chronic diarrhea or malabsorption; pre-existent progressive neuromuscular disease, and Metastatic cancer
4. Pregnancy and breast feeding
5. Medications: immunosuppressive chemotherapy; regular use of digoxin, amiodarone, verapamil or protease inhibitors.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2021-10-30 (Actual)

PRIMARY OUTCOMES:
- To assess the percentage of cure of the patients | up to 14 days
  evauated by normalization of clinical evaluation, laboratory investigations, and imaging
- Study the time to recovery | up to 14 days
  Evaluated by stay days in hospital

SECONDARY OUTCOMES:
- to assess side effects seen during the trial | up to 14 days
  assessed according clinical evaluation and the appropriate laboratory investigation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed S Abdulamir, MD, Study Chair — Alnahrin University
Locations (1):
- University of Baghdad, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No